CLINICAL TRIAL: NCT04353635
Title: The Assessment of Prediction of Soft Tissue Changes Following the Surgical Correction of Dento-facial Deformities Using Dolphin 3D Software Package.
Brief Title: Prediction Accuracy of Dolphin 3D in Bimax Surgery for Class III
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Principal Investigator, Nehal Ibrahim Ahmed Shobair, Key Investigator, Ain Shams University
Other Study IDs: 732092017
Record Dates: First submitted 2020-03-29; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Orthognathic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with class III dentofacial deformity: No intervention as it will be a retrospective study
  Interventions: Device: dolphin 3d

INTERVENTIONS:
Device: dolphin 3d — software

SUMMARY:
Patients with class III dentofacial deformity who are in need of surgical correction are now able to see the potential changes to their faces before the actual operation. Dolphin 3d is one of the few software packages that is used for orthognathic planning and prediction of soft tissue changes. The direct effect of the prediction procedure over patient's and surgeon decisions makes it important to guarantee a high level of accuracy of operational results prediction. This study is designed to investigate the accuracy of Dolphin 3d software for the prediction of postoperative soft tissue changes following specific surgical procedure which is the combined maxillary advancement and mandibular setback, commonly used for correction of class III facial deformity cases. The study data will be collecting retrospectively. The difference between the pre-operative soft tissue prediction and the 6-month postoperative results will be analysed. The results of this study will help to determine whether this software package is accurate enough to be considered as a surgical assistance tool helping both surgeons and patients in treatment planning and decision-making procedure respectively.

DETAILED DESCRIPTION:
The study will employ the pre-existing CBCT images routinely captured for orthognathic surgery patients in Glasgow dental hospital and school.

The CBCT scans of class III patients who undergone maxillary advancement with minimal or without impaction and mandibular setback will be identified.

The preoperative and 6 months postoperative CBCT images will be anonymised The surgical planning and soft tissue prediction will be performed on the preoperative images using Dolphin3d software.

The resultant soft tissue 3D model will be superimposed on the actual postoperative soft tissue model.

Analysis of the difference between the prediction and the actual postoperative will be performed to quantify the difference between them in order to assess the accuracy of the software prediction.

The sample will be collected according to the inclusion and exclusion criteria. Pre and post operation CBCT voxel based super imposition using ONDEMAND 3d. The surgical movement will be quantified using direct slice land-marking . Using the pre-operattion CBCT to do the surgical mock up and the soft tissue simulation on dolphin 3D.

Segment the soft tissue of the prediction. Soft tissue surface models of the simulation and the actual postoperative images were generated and exported as STLs.

Generic meshes conformation dense correspondence analysis. Superimposition of the predicted and the post operative STLs. Using VR mesh software, the mesh will be segmented into pre-identified anatomical regions.

The distance between the corresponding vertices will be displayed as a colour scale in milli-meter and will be analysed in the individual dimension of space (x, y and z) using in-house software and each dimension will be displayed as a colour coded distance map.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have class III facial deformity to be corrected using bimaxillary orthognathic surgery.
2. No medical problems that might interfere with general anesthesia or interfere with bone and soft tissue healing.

Exclusion Criteria:

1. There are craniofacial anomalies including cleft lip/palate,
2. Patient have previous maxillofacial operations or facial scars,
3. Correction mandates multi-segment Le Fort I osteotomies,
4. There are orthodontic appliances in place at the time of T1 records.
5. Genioplasty is recommended for deformity correction.
6. There is facial Asymmetry.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with classIII dentofacial deformity
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
The difference between prediction and actual postoperative | 6 months
  The difference between prediction and actual postoperative. The distance between the corresponding vertices will be displayed as a colour scale in milli-meter and will be analysed in the individual dimension of space (x, y and z) using in-house software and each dimension will be displayed as a colour coded distance map.

SECONDARY OUTCOMES:
The distance between the corresponding vertices | 6 months
  Tthe secondary outcome measures will be the distance between the corresponding vertices which will be displayed as a colour scale in milli-meters

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT04353635/Prot_SAP_000.pdf